CLINICAL TRIAL: NCT05237518
Title: Accuracy Evaluation of EarlySense Device, a Smaller Shape Sensor With BLE Connection to Processing Unit (HUB)) for Use While Two People Are in Bed ("Home Use" Scenario)
Brief Title: Accuracy Evaluation of EarlySense With Modified Sensor (Smaller Shape Sensor With BLE) at Home Setting Monitoring a Subject While Partner in Bed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: EarlySense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ES-CLC-2022-001
Record Dates: First submitted 2022-01-13; First posted 2022-02-14 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-02

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 36 adults (Other): The test group should include both men and women subjects. Two equal sizes (18) sub-groups will be enrolled such that each sub-group will be monitored while lying on a different mattress type.
  Interventions: Device: EarlySense Noomi system

INTERVENTIONS:
Device: EarlySense Noomi system — The EarlySense device is intended for continuous contact-free monitoring of heart rate and respiration rate at home, or in professional healthcare settings. The system is intended for remote monitoring of patients by healthcare professionals and is indicated mainly for elderly population monitoring.
  Other Names: EarlySense™ device

SUMMARY:
Accuracy evaluation of EarlySense device, a smaller shape sensor with BLE connection to processing unit (HUB)) for use while two people are in bed ("Home Use" scenario) The EarlySense device is intended for continuous contact-free monitoring of heart rate and respiration rate at home, or in professional healthcare settings. The system is intended for remote monitoring of patients by healthcare professionals and is indicated mainly for elderly population monitoring.

The modified version of this product which is the subject of this validation study allows monitoring of subjects when there is a second person in the same bed ("Home scenario" environment). The objective of this study is to evaluate the accuracy of the device in determining Respiration Rate (Br./min) and Heart Rate (BPM) at home environment, while two people are in the same double bed. The study aims to demonstrate that partner presence doesn't affect the monitoring accuracy of the subject that is being measured.

The continuous monitoring will last for duration of 90 minutes for each subject, unless the participant requests termination of the experiment or as per the physician's instructions. Subjects admitted to the study will be monitored using both Capnography and ECG- as reference devices. The EarlySense revised sensor will be placed under one of the two-mattress types incorporated into the study. Both mattresses are typical double bed mattresses of 160 X 200 cm with two different internal structure composition. The sensor will be placed directly below the subject's thorax area on one of the mattress sides. The signals collected by the sensor will be communicated via BLE to the processing unit (HUB).

Following connecting the subject to the reference devices, both the subject and the partner will be instructed on the actions they should perform through the stages of the experiment.

The subject will lie on the mattress side where the EarlySense sensor is located, while the partner will be instructed to enter the other side of the mattress. At this time, the experiment will start, and the clock will start running.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Sleeping with a partner in bed
* Willing to sign the consent form

Exclusion Criteria:

* Subjects with arrhythmia will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Respiration Rate (Br./min) | 90 minutes
  Measurement obtained from study device will be compared to measurement obtained from SOC device.
Heart Rate (BPM) | 90 minutes
  Measurement obtained from study device will be compared to measurement obtained from SOC device.